CLINICAL TRIAL: NCT05273801
Title: Assessing Feasibility, Efficacy, and Acceptability of Visual Feedback During HR Monitoring in Rehabilitation
Brief Title: Assessing Visual Feedback of HR Monitoring in Rehabilitation - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Miriam Rafferty, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00216223
Record Dates: First submitted 2022-02-01; First posted 2022-03-10 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Exercise Therapy; Heart Rate Determination
Keywords: Hospitals, Rehabilitation; Exercise Therapy; Heart Rate Determination; Rehabilitation Centers

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in a single arm where they may receive HR monitoring with visual feedback or HR monitoring with no visual feedback. Observed condition will alternate by session.
Masking Description: All individuals involved in the study will be aware when HR feedback as well as monitoring occurs during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational HR monitoring (Experimental): Participants will receive 2 intervention conditions: HR monitoring with visual feedback, and HR monitoring without visual feedback. Observed condition will alternate by session. The investigators will monitor overall HR response, mean time HR and time in target zone, Rate of perceived exertion (RPE), and provider behavior to HR monitoring prior to HR monitoring, with visual feedback and without visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a television (TV) monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
  Interventions: Device: Heart Rate Recording from Multiple Participants, No Visual Feedback; Device: Visual Feedback of Multiple Participant Heart Rates

INTERVENTIONS:
Device: Heart Rate Recording from Multiple Participants, No Visual Feedback — Heart rates are recorded from multiple participants during the group sessions. However during this intervention, it will not be cast to a TV for feedback to the participant or clinician.
  Other Names: Heart Zones, Inc
Device: Visual Feedback of Multiple Participant Heart Rates — Visual feedback of HR is provided through a TV monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
  Other Names: Heart Zones, Inc

SUMMARY:
Monitoring heart rate during exercise can provide feedback to the patient and provider that the patient is exercising in the appropriate, individualized and safe range for them. This is particularly important in a group setting when multiple individuals are supervised by one provider. This study is interested in assessing the difference in intensity of care delivered when visual feedback of heart rate is provided compared to no visual feedback of heart rate in rehabilitation. Visual feedback of heart rate will be provided through Heart Zones, a platform which synthesizes multiple signals from externally worn heart rate monitors. This study is interested in better understanding the acceptability, feasibility and appropriateness of this technology when used in rehabilitation.

DETAILED DESCRIPTION:
OBJECTIVES:

The purpose of this investigation is to determine if knowledge of heart rate (HR) and target HR zones (HRzone), with visual feedback vs no feedback of HR or HRzone improves patient exercise intensity during rehabilitation. The central hypothesis for this study is with visual feedback of HR and target HR zones with instruction about exercise intensity and targets will increase patient HR intensity during sessions within a safe range set by their medical team. For purposes of this study, patients will be monitored in inpatient sessions and is inclusive of all individuals with chronic health conditions. Physical activity and exercise guidelines recommend everyone, including those with chronic health conditions, strive for 150 minutes of moderate intensity aerobic exercise per week. This study will contribute to the knowledge of how patients achieve recommended individual HR and moderate-high intensity zones during exercise.

Aim 1: Measure the extent to which monitoring and education regarding intensity is provided (1) when providers know HR monitoring is occurring but without visual feedback for the group, and (2) with visual feedback of HR monitoring in a group setting.

The investigators hypothesize providers will modify their behavior in the number of times they ask about intensity, adjust session intensity or provide education regarding intensity when visual feedback is provided compared to no feedback.

Aim 2: Determine the safety of using Heart Zones technology in rehabilitation settings for increasing participant exercise intensity.

The investigators hypothesize the technology will be safe without an increase in number of adverse events throughout their rehabilitation stay.

Aim 3: Assess patient acceptability, exercise self-efficacy and confidence following use of Heart Zones technology in group settings.

The investigators hypothesize use of Heart Zones technology in rehabilitation with feedback will increase participant self-efficacy and confidence in reaching higher exercise intensities, and will be well accepted.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to inpatient rehabilitation, day rehabilitation or participant in community fitness
* Qualifies for group therapy based on diagnosis and insurance reimbursement
* Physician clearance for participation

Exclusion Criteria:

* Unable to provide informed consent due to cognitive impairment
* Inability to communicate with investigators
* Sternal Precautions
* Individuals with Left Ventricular assist devices
* Pregnant women
* Uncontrolled Hypertension
* Serious and unstable cardiac arrhythmias
* Loss of bilateral upper extremity sensation
* At high risk for skin breakdown due to poor skin integrity (open wound, fragile skin, etc)
* Previous participation in this study while in another level of care in the last 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Rafferty, DPT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Pilot data of individuals clinical care with plan for future work to validate process.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 of 18 participants were included. One participant did not meet inclusion criteria. Observed providers were not consented to the study so were not considered enrolled
Groups:
- Observational HR Monitoring: Participants were observed in 2 conditions: 1) HR monitoring without visual feedback and 2) HR monitoring with visual feedback. The investigators will monitor overall HR response, mean time HR and time in target zone, rate of perceived exertion (RPE), and provider behavior to HR monitoring with visual feedback and without visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a television (TV) monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
Period: Overall Study
Arm/Group | Observational HR Monitoring
Started | 18
Number of Participants Who Recieved HR Monitoring Without Visual Feedback | 15
Number of Participants Who Received HR Monitoring With Visual Feedback | 15
Completed | 17
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Only one arm is described because the same unique participants participated in 2 conditions (HR monitoring with visual feedback, HR monitoring without visual feedback), however not in a formal structured crossover design to allow separation. One arm is required for accurate demographic reporting (n total 18 consented, 17 participants at baseline). Providers were not consented to the study so were not considered enrolled.
Groups:
- Observational HR Monitoring: Participants were observed in 2 conditions: 1) HR monitoring without visual feedback and 2) HR monitoring with visual feedback. The investigators will monitor overall HR response, mean time HR and time in target zone, RPE, and clinician behavior to HR monitoring prior to HR monitoring, with visual feedback and without visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a TV monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
Arm/Group | Observational HR Monitoring
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants on Beta Blocker Medications [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Provider Behavior
Description: Number of times heart rate (beats/minute), Rate of perceived exertion (6-20, higher = greater perceived exertion) or intensity (asked in session by HR/RPE) is monitored and/or modified based on feedback during rehabilitation sessions.
Time Frame: Through study completion, an average of 3 months
Population: Participants are part of one arm and may have been observed in either of these assigned interventions. For clarity, assigned intervention are separated into "arms". Participants analyzed in each intervention group are <17 because not all participants received each intervention due to medical care (unexpected discharge, transfer to acute hospital, schedule). Providers were not consented to the study so were not considered enrolled. Provider Behavior data were not collected from providers.
Measure: Mean (Standard Deviation); unit: observations
Units Other Than Participants: session count
Groups:
- HR Monitor, no Visual Feedback: Participants will have HR monitoring in their group sessions where visual feedback is not provided. The investigators will monitor overall HR response, mean HR and time in target HR zone, RPE and clinician behavior to HR monitor on patient during these sessions.
  Heart Rate Recording from Multiple Participants, No visual feedback: Heart rates are recorded from multiple participants during the group sessions. However during this intervention, it will not be cast to a TV for feedback to the participant or clinician. Participants listed is number of sessions observed.
- HR Monitor, With Feedback: Participants will have HR monitoring with visual feedback during group sessions. The investigators will monitor overall HR response, mean time HR and time in target zone, RPE, and clinician behavior to HR monitoring with visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a TV monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity. Participants listed is number of sessions observed.
Arm/Group | HR Monitor, no Visual Feedback | HR Monitor, With Feedback
Number analyzed (Participants) | 15 | 15
Number analyzed (session count) | 31 | 28
observations
  How frequently provider ask about RPE/HR during session | 0.38 (0.97) | 0.48 (0.90)
  How frequently education provided regarding HR/RPE during session | 0.62 (1.24) | 1.43 (1.47)
  How frequently HR/RPE target is mentioned in session | 0.33 (1.11) | 4.91 (7.38)
  How frequently provider modifies session/task to reach HR/RPE target | 0.29 (0.64) | 2.17 (2.87)
  How frequently providers monitor HR/RPE during session | 5.14 (8.70) | 20.43 (12.09)
Statistical Analysis 1: Comparison: HR Monitor, no Visual Feedback vs HR Monitor, With Feedback; How frequently clinician ask about RPE/HR during session; Test type: Superiority; p = 0.73, t-test, 2 sided
Statistical Analysis 2: Comparison: HR Monitor, no Visual Feedback vs HR Monitor, With Feedback; How frequently education provided regarding HR/RPE during session; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: HR Monitor, no Visual Feedback vs HR Monitor, With Feedback; How frequently HR/RPE target is mentioned in session; Test type: Superiority; p = 0.007, t-test, 2 sided
Statistical Analysis 4: Comparison: HR Monitor, no Visual Feedback vs HR Monitor, With Feedback; How frequently clinician modifies session/task to reach HR/RPE target; Test type: Superiority; p = 0.005, t-test, 2 sided
Statistical Analysis 5: Comparison: HR Monitor, no Visual Feedback vs HR Monitor, With Feedback; How frequently clinicians monitor HR/RPE during session; Test type: Superiority; p = 0.00001, t-test, 2 sided

2. Secondary Outcome: Patient Participant Self-Efficacy and Confidence
Description: Using a scale from 0-100% (higher is better), participant's rate their self-efficacy and confidence in their ability to achieve target exercise intensity and confidence in performing the activity without a heart rate monitor after each session. Data from each session are averaged to create a single value per participant.
Time Frame: Assessed during therapy sessions (1-4 hrs/day, up to 5 days per week) through the duration of patient's rehabilitation stay (approximately 5-60 days).
Population: Participants are part of one arm and may have been observed in either of these assigned interventions. For clarity, assigned intervention are separated into "arms". Participants analyzed in each intervention group are <17 because not all participants received each intervention due to medical care (unexpected discharge, transfer to acute hospital, schedule). Providers were not consented to the study so were not considered enrolled.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HR Monitor, no Feedback: Participants will have HR monitoring in their group sessions where visual feedback is not provided. The investigators will monitor overall HR response, mean HR and time in target HR zone, RPE and clinician behavior to HR monitor on patient during these sessions.
  Heart Rate Recording from Multiple Participants, No visual feedback: Heart rates are recorded from multiple participants during the group sessions. However during this intervention, it will not be cast to a TV for feedback to the participant or clinician.
- HR Monitor, With Feedback: Participants will have HR monitoring with visual feedback during group sessions. The investigators will monitor overall HR response, mean time HR and time in target zone, RPE, and clinician behavior to HR monitoring with visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a TV monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
Arm/Group | HR Monitor, no Feedback | HR Monitor, With Feedback
Number analyzed (Participants) | 15 | 15
score on a scale
  Patient self-confidence (0-100%) reaching target intensity in session. | 72.9 (25.9) | 77.5 (24.3)
  Patient self-rating of confidence to continue to reach target without HR monitor in future (0-100%) | 85.0 (19.2) | 79.3 (20.4)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months
Description: Adverse event collection occurred at end of each data collection session. The number of participants potentially at risk is <17 because not all participants received each intervention due to medical care (unexpected discharge, transfer to acute hospital, schedule). Providers were not consented to the study so were not considered enrolled.
Groups:
- HR Monitor, no Feedback: Participants will have HR monitoring in their group sessions where visual feedback is not provided during group session. The investigators will monitor overall HR response, mean HR and time in target HR zone, RPE and provider behavior to HR monitor on patient during these sessions.
  Heart Rate Recording from Multiple Participants, No visual feedback: Heart rates are recorded from multiple participants during the group sessions. However during this intervention, it will not be cast to a TV for feedback to the participant or clinician.
- HR Monitor, With Feedback: Participants will have HR monitoring with visual feedback during group sessions. The investigators will monitor overall HR response, mean time HR and time in target zone, RPE, and provider behavior to HR monitoring with visual feedback.
  Visual Feedback of Multiple Participant Heart Rates: Visual feedback of HR is provided through a TV monitor. Multiple heart rates can be displayed and recorded simultaneously allowing for group encouragement, continuous monitoring and adjustment of all participants to ensure reaching appropriate target intensity.
Arm/Group | HR Monitor, no Feedback | HR Monitor, With Feedback
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Heart rate data collected from multiple brands of devices due to readability issue in some patients. Some patients' peripheral circulation and use of devices affected HR transmission; thus possibly affecting reliability and consistency of heart rate data collected in sessions. Given this, clinician's behavior may have been affected when providing visual feedback. This data served as pilot exploratory data for future work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT05273801/Prot_SAP_000.pdf